CLINICAL TRIAL: NCT00702520
Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established After Controlled Ovarian Stimulation in Clinical Trial 38833 for Org 36286 (Corifollitropin Alfa)
Brief Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established in Clinical Trial 38833 (P05783)
Acronym: Care
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05783; 38834 (Other: Organon); MK-8962-010 (Other: Merck); 2005-000062-40 (EudraCT Number)
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy; Neonates
Keywords: Neonatal outcome; Congenital malformations; In-Vitro fertilization; Controlled ovarian stimulation; Follow-up
MeSH Terms: conditions — Congenital Abnormalities | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; Triptorelin Pamoate; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Corifollitropin alpha 100 ug: In the base study (P05788, 38833, NCT00702351), participants were pre-treated with daily subcutaneous (SC) injections of 0.1 mg triptorelin started between Day 21 and 24 of the menstrual cycle (mid luteal phase). After suppression of endogenous luteinizing hormone (LH) and follicle stimulating hormone (FSH) was confirmed by estradiol (E2) and progesterone (P) measurements, a single dose of corifollitropin alpha 100 μg was administered in participants weighing <= 60 kg. From stimulation Day 8 onwards, treatment was continued with daily SC of recombinant follicle stimulating hormone (recFSH) injections (maximally 200 IU) up to and including the day of administration of human chorionic gonadotprophin (hCG). No study medications were administered in the present P05783 study (38834, NCT00702520).
  Interventions: Drug: Corifollitropin alpha (MK-8962, Org 36286) 100 ug; Drug: Triptorelin; Biological: Recombinant follicle stimulating hormone (recFSH); Biological: Human chorionic gonadotprophin (hCG).
- Corifollitropin alpha 150 ug: In the base study (P05788, 38833, NCT00702351), participants were pre-treated with daily SC injections of 0.1 mg triptorelin started between Day 21 and 24 of the menstrual cycle (mid luteal phase). After suppression of endogenous LH and FSH was confirmed by E2 and P measurements, a single dose of corifollitropin alpha 150 μg was administered in participants weighing >= 50 kg. From stimulation Day 8 onwards, treatment was continued with daily SC of recFSH injections (maximally 200 IU) up to and including the day of administration of hCG. No study medications were administered in the present P05783 study (38834, NCT00702520).
  Interventions: Drug: Corifollitropin alpha (MK-8962, Org 36286) 150 ug; Drug: Triptorelin; Biological: Recombinant follicle stimulating hormone (recFSH); Biological: Human chorionic gonadotprophin (hCG).

INTERVENTIONS:
Drug: Corifollitropin alpha (MK-8962, Org 36286) 100 ug — Subcutaneous administration of corifollitropin alpha at a dose of 100 ug
  Groups: Corifollitropin alpha 100 ug
Drug: Corifollitropin alpha (MK-8962, Org 36286) 150 ug — Subcutaneous administration of corifollitropin alpha at a dose of 150 ug
  Groups: Corifollitropin alpha 150 ug
Drug: Triptorelin — Daily SC injections of 0.1 mg triptorelin started between Day 21 and 24 of the menstrual cycle (mid luteal phase).
Biological: Recombinant follicle stimulating hormone (recFSH) — From stimulation Day 8 onwards, treatment was continued with daily SC of recFSH injections (maximally 200 IU) up to and including the day of administration of hCG.
Biological: Human chorionic gonadotprophin (hCG). — HCG was administered as a single subcutaneous injection of 5,000 to 10,000 international units.

SUMMARY:
The objective of this trial is to evaluate whether corifollitropin alfa (MK-8962, Org 36286) treatment for the induction of multifollicular growth in women undergoing Controlled Ovarian Stimulation (COS) prior to in vitro fertilization (IVF) or Intracytoplasmic Sperm Injection (ICSI) is safe for pregnant participants and their offspring.

DETAILED DESCRIPTION:
This is a follow-up protocol to prospectively monitor pregnancy, delivery, and neonatal outcomes of all women who were treated with corifollitropin alfa and became pregnant during the base Trial 38833. For this follow-up trial (38834), no investigational products will be administered and no study specific assessments are required, but information will be obtained as per standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants who received one dose of corifollitropin alfa in Trial 38833;
* Ongoing pregnancy confirmed by ultrasound at least 10 weeks after embryo transfer in Trial 38833;
* Able and willing to give written informed consent.

Exclusion Criteria:

* None

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with an ongoing pregnancy at least 10 weeks after embryo transfer in Trial 38833 were enrolled in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2007-11-07 (Actual); Study Completion 2008-01-15 (Actual)

REFERENCES:
- [Derived] Bonduelle M, Mannaerts B, Leader A, Bergh C, Passier D, Devroey P. Prospective follow-up of 838 fetuses conceived after ovarian stimulation with corifollitropin alfa: comparative and overall neonatal outcome. Hum Reprod. 2012 Jul;27(7):2177-85. doi: 10.1093/humrep/des156. Epub 2012 May 15. PMID 22587997

RESULTS

PARTICIPANT FLOW:
Groups:
- Expectant Mothers Administered Corifollitropin Alpha 100 ug: In the base study (P05788, 38833, NCT00702351), after suppression of endogenous LH and FSH was confirmed by E2 and P measurements, a single dose of corifollitropin alpha 100 μg was administered in participants weighing <= 60 kg. No study medications were administered in the follow-up P05783 study.
- Expectant Mothers Administered Corifollitropin Alpha 150 ug: In the base study (P05788, 38833, NCT00702351), after suppression of endogenous LH and FSH was confirmed by E2 and P measurements, a single dose of corifollitropin alpha 150 μg was administered in participants weighing >= 50 kg. No study medications were administered in the follow-up P05783 study.
- Infants From Mothers Administered Corifollitropin Alpha 100 ug: Infants born to mothers who received 100 ug corifollitropin alfa in the base study (P05788, 38833, NCT00702351), were followed for safety and efficacy in the current follow-up study (P05783, 38834, NCT00702520). No study medications were administered in the follow-up P05783 study.
- Infants From Mothers Administered Cori. Alpha 150 ug: Infants from mothers who received 150 ug corifollitropin alfa in the base study (P05788, 38833, NCT00702351), were followed for safety and efficacy in the current follow-up study (P05783, 38834, NCT00702520). No study medications were administered in the follow-up P05783 study.
Period: Base Study P05788 - Assigned Treatment
Arm/Group | Expectant Mothers Administered Corifollitropin Alpha 100 ug | Expectant Mothers Administered Corifollitropin Alpha 150 ug | Infants From Mothers Administered Corifollitropin Alpha 100 ug | Infants From Mothers Administered Cori. Alpha 150 ug
Started | 25 | 25 | 0 | 0
Treated With Corifollitropin Alpha | 25 | 24 | 0 | 0
Treated With hCG and Had Oocyte Pick-up | 25 | 24 | 0 | 0
Completed | 25 | 24 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Spontaneous pregnancy | 0 | 1 | 0 | 0
Period: Base Study P05788 - Embryo Transfer
Arm/Group | Expectant Mothers Administered Corifollitropin Alpha 100 ug | Expectant Mothers Administered Corifollitropin Alpha 150 ug | Infants From Mothers Administered Corifollitropin Alpha 100 ug | Infants From Mothers Administered Cori. Alpha 150 ug
Started | 25 | 24 | 0 | 0
Embryo Transfer | 22 | 18 | 0 | 0
Completed | 22 | 18 | 0 | 0
Not Completed | 3 | 6 | 0 | 0
Not completed — No embryo transfer | 3 | 6 | 0 | 0
Period: Base Study P05788 - Follow-Up
Arm/Group | Expectant Mothers Administered Corifollitropin Alpha 100 ug | Expectant Mothers Administered Corifollitropin Alpha 150 ug | Infants From Mothers Administered Corifollitropin Alpha 100 ug | Infants From Mothers Administered Cori. Alpha 150 ug
Started | 22 | 18 | 0 | 0
Ongoing Pregnancy at 10 Weeks | 7 | 8 | 0 | 0
Completed | 7 | 8 | 0 | 0
Not Completed | 15 | 10 | 0 | 0
Not completed — No ongoing pregnancy at 10 weeks | 15 | 10 | 0 | 0
Period: Follow-up Study P05783
Arm/Group | Expectant Mothers Administered Corifollitropin Alpha 100 ug | Expectant Mothers Administered Corifollitropin Alpha 150 ug | Infants From Mothers Administered Corifollitropin Alpha 100 ug | Infants From Mothers Administered Cori. Alpha 150 ug
Started | 7 | 8 | 8 (This is the number of infants born from mothers administered Corifollitropin alpha 100 ug.) | 11 (This is the number of infants born from mothers administered Corifollitropin alpha 150 ug.)
Completed | 7 | 8 | 8 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants reflects the number of participants that started the P05783 follow-up study and not the number of participants in the P05788 base study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Expectant Mothers Administered Corifollitropin Alpha 100 ug | Expectant Mothers Administered Corifollitropin Alpha 150 ug | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.1 (2.0) | 31.3 (4.2) | 30.7 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Expectant Mothers Experiencing Adverse Events (AEs)
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the study drug.
Time Frame: Up to 1 Year
Population: Follow-up safety analysis was performed on expectant mothers who received corifollitropin alfa in the base study P05690 (NCT00702845) and who enrolled in the follow-up study (P05783, 38834, NCT00702520).
Measure: Number; unit: Participants
Arm/Group | Expectant Mothers Administered Corifollitropin Alpha 100 ug | Expectant Mothers Administered Corifollitropin Alpha 150 ug
Number analyzed (Participants) | 7 | 8
Participants | 7 | 6

2. Primary Outcome: Number of Expectant Mothers Experiencing Serious AEs (SAEs)
Description: An AE or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Up to 1 Year
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Expectant Mothers Administered Corifollitropin Alpha 100 ug | Expectant Mothers Administered Corifollitropin Alpha 150 ug
Number analyzed (Participants) | 7 | 8
Participants | 2 | 2

3. Primary Outcome: Number of Infants Experiencing AEs
Description: as for outcome 1
Time Frame: Up to 1 Year
Population: Follow-up safety analysis was performed on live born infants delivered by expectant mothers who received corifollitropin alfa in the base study P05690 (NCT00702845) and who enrolled in the follow-up study (P05783, 38834, NCT00702520).
Measure: Number; unit: Participants
Arm/Group | Infants From Mothers Administered Corifollitropin Alpha 100 ug | Infants From Mothers Administered Cori. Alpha 150 ug
Number analyzed (Participants) | 8 | 11
Participants | 6 | 11

4. Primary Outcome: Number of Infants Experiencing SAEs
Description: as for outcome 2
Time Frame: Up to 1 Year
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Infants From Mothers Administered Corifollitropin Alpha 100 ug | Infants From Mothers Administered Cori. Alpha 150 ug
Number analyzed (Participants) | 8 | 11
Participants | 6 | 7

5. Primary Outcome: Take-Home Baby Rate
Description: The take-home baby rate was calculated as the number of participants with a least one live born infant in the follow-up study (P05783, 38834, NCT00702520) relative to the number of participants treated with Corifollitropin alpha in the base study (P05788, 38833, NCT00702351).
Time Frame: Birth of a one or more live babies (Up to 1 year)
Population: Participants treated with Corifollitropin alpha in the base study (P05788, 38833).
Measure: Number; unit: Percentage of participants
Arm/Group | Expectant Mothers Administered Corifollitropin Alpha 100 ug | Expectant Mothers Administered Corifollitropin Alpha 150 ug
Number analyzed (Participants) | 25 | 24
Percentage of participants | 28.0 | 33.3

ADVERSE EVENTS:
Time Frame: Up to 1 year
Groups:
- Expectant Mothers Administered Corifollitropin Alpha 100 ug: In the base study (P05788, 38833, NCT00702351), after suppression of endogenous LH and FSH was confirmed by E2 and P measurements, a single dose of corifollitropin alpha 100 μg was administered in participants weighing <= 60 kg. No study medications were administered in the P05783 study (38834, NCT00702520).
- Fetuses/Infants From Mothers Administered Cori. Alpha 100 ug: Fetuses/Infants from mothers who received 100 ug corifollitropin alfa in the base study (P05788, 38833, NCT00702351), were followed for safety and efficacy in the current follow-up study (P05783, 38834, NCT00702520) according to standard practice. No study medications were administered in the follow-up P05783 study.
- Fetuses/Infants From Mothers Administered Cori. Alpha 150 ug: Fetuses/Infants from mothers who received 150 ug corifollitropin alfa in the base study (P05788, 38833, NCT00702351), were followed for safety and efficacy in the current follow-up study (P05783, 38834, NCT00702520) according to standard practice. No study medications were administered in the follow-up P05783 study.
Arm/Group | Expectant Mothers Administered Corifollitropin Alpha 100 ug | Expectant Mothers Administered Corifollitropin Alpha 150 ug | Fetuses/Infants From Mothers Administered Cori. Alpha 100 ug | Fetuses/Infants From Mothers Administered Cori. Alpha 150 ug
Serious Adverse Events (participants affected / at risk) | 2/7 | 2/8 | 6/8 | 7/11
Other Adverse Events (participants affected / at risk) | 7/7 | 6/8 | 5/8 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Expectant Mothers Administered Corifollitropin Alpha 100 ug (N=7) | Expectant Mothers Administered Corifollitropin Alpha 150 ug (N=8) | Fetuses/Infants From Mothers Administered Cori. Alpha 100 ug (N=8) | Fetuses/Infants From Mothers Administered Cori. Alpha 150 ug (N=11)
Accessory auricle (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital choroid plexus cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital labia pudendi adhesions (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital laryngeal stridor (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital naevus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pilonidal cyst congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pulmonary valve stenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scaphocephaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skull malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholestasis of pregnancy (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intercostal retraction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal anoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Expectant Mothers Administered Corifollitropin Alpha 100 ug (N=7) | Expectant Mothers Administered Corifollitropin Alpha 150 ug (N=8) | Fetuses/Infants From Mothers Administered Cori. Alpha 100 ug (N=8) | Fetuses/Infants From Mothers Administered Cori. Alpha 150 ug (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Craniotabes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Fever neonatal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suprapubic pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal identification test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intrapartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal laceration (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Placenta praevia haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infantile apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervix cerclage procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine dilation and curettage (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor recognizes the right of the investigator(s) to publish, but all publications must be based on data validated and released by the sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial described in this protocol will first be submitted to the sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.